CLINICAL TRIAL: NCT05146063
Title: LNK Participates in Insulin Resistance in Polycystic Ovary Syndrome by Regulating Adipose Glucose Transport
Brief Title: LNK in Polycystic Ovary Syndrome With Insulin Resistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2021-187
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Polycystic Ovarian Syndrome; Insulin Resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycystic ovary syndrome patients with insulin resistance
  Interventions: Diagnostic Test: Take the patient's subcutaneous fat tissue to detect the expression of LNK
- Polycystic ovary syndrome patients without insulin resistance
  Interventions: Diagnostic Test: Take the patient's subcutaneous fat tissue to detect the expression of LNK

INTERVENTIONS:
Diagnostic Test: Take the patient's subcutaneous fat tissue to detect the expression of LNK — Take the patient's subcutaneous fat tissue to detect the mRNA and protein expression levels of LNK by RT-qPCR and western blot.

SUMMARY:
Insulin resistance (IR) is an important pathological feature of polycystic ovary syndrome (PCOS), with an incidence rate of up to 85%, which seriously affects the patient's fertility, quality of life, and offspring health, but the mechanism is unknown. The adaptor protein LNK is closely related to metabolic diseases. Our exome sequencing has found that the mutation rate of LNK gene in patients with PCOS and IR is high. Studies have found that LNK can affect adipose inflammation and impair glucose tolerance. Whether LNK is related to fat metabolism is worth further study. Our previous research found that: LNK expression was significantly increased in adipose tissue of patients with PCOS and IR. Knockout of LNK in PCOS IR model mice can reduce serum triglycerides, free fatty acids, high-sensitivity C-reactive protein levels and reduce fatty liver occurrence, which indicates that LNK has a mitigating effect on IR. Mechanism studies have shown that LNK knockout can upregulate the glucose transporter Glut4, also LNK and insulin receptor substrate IRS-1 can form protein complexes. Based on the above research basis, we propose the following scientific hypothesis: LNK in adipose tissue can regulate insulin signaling pathway by binding to IRS-1, downregulate Glut4, and participate in PCOS IR occurrence. This project intends to clarify the specific mechanism by which LNK regulates glucose transport and participate in IR in combination with clinical specimens, animal models and cell experiments, and provide scientific basis for LNK as a potential therapeutic target for PCOS IR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with polycystic ovary syndrome who meet the 2003 Rotterdam criteria

Exclusion Criteria:

* Do not meet the diagnostic criteria for polycystic ovary syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with polycystic ovary syndrome who met the 2003 Rotterdam criteria were divided into insulin resistance group and non-insulin resistance group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mRNA expression levels of LNK | 2 years
  The expression level of LNK mRNA in the subcutaneous adipose tissue of the PCOS patients
protein expression levels of LNK | 2 years
  The expression level of LNK protein in the subcutaneous adipose tissue of the PCOS patients

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Study Director — Sun Yat-sen Memorial Hospital, Sun Yat-sen Univers
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided